CLINICAL TRIAL: NCT02853942
Title: The Research of Autologous Adipose Mesenchymal Stem Cell Transplantation for Treatment of Facial 、Auditory Nerve Dysfunction of Patients With Hemifacial Spasm After Microvascular Decompression.
Brief Title: Autologous Adipose Mesenchymal Stem Cell Transplantation in the Treatment of Patients With Hemifacial Spasm
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Shiting Li, Office of clinical research of Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-16-012
Record Dates: First submitted 2016-07-14; First posted 2016-08-03 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Injury of Facial Nerve, Unspecified Side, Initial Encounter
MeSH Terms: conditions — Facial Nerve Injuries | interventions — mecobalamin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stem cell therapy group (Experimental): Using the international standard 14G (diameter 1.54mm) needle inject autologous adipose derived mesenchymal stem cells 2ml to facial nerve, the effective release of the concentration is 100 million stem cells / ml.
  Interventions: Biological: Autologous adipose stem cell therapy; Drug: Mecobalamin
- Neurotrophic drugs treatment group (Experimental): Patients were treated with routine drug therapy，do not inject stem cell to the facial nerve of patient
  Interventions: Drug: Mecobalamin

INTERVENTIONS:
Biological: Autologous adipose stem cell therapy
  Arms: Stem cell therapy group
Drug: Mecobalamin

SUMMARY:
Main purpose：In the face of listening to nerve injury at early stage, utilizing autologous adipose stem cell transplantation in the treatment of makes the acceptance micro vascular decompression hemifacial spasm patients to nerve function to obtain a better recovery.

Secondary purpose ：To clarify the efficacy of stem cells in the treatment of cranial nerve dysfunction, and to provide evidence for the treatment of other cranial nerve dysfunction.

Cases in group：Appearing on the surface of microvascular decompression for hemifacial spasm to decrease neural electrophysiological index of patients research design：Single center, prospective, randomized, double-blind, controlled Observation index：Facial nerve clinical score, facial nerve muscle compound action potential, electrical measurement, cerebrospinal fluid index Evaluation of therapeutic effect：Facial nerve function evaluation (House-Brackmann classification, facial nerve function classification scale SFGS), facial nerve electrophysiology evaluation (facial nerve muscle compound action potential), electric measurement Safety evaluation：Clear evaluation of hemifacial spasm and micro vascular decompression were listening to nerve in intracranial segment wrapped around the autologous fat stem cell therapy overall safety and evaluation methods including adverse events, laboratory tests, vital signs, electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

1. the age of 18 ~ 80 years old;
2. no surgical contraindications, accept facial nerve microvascular decompression surgery;
3. to enter into the group's informed consent and sign the consent form for clinical research.
4. patients with preoperative facial nerve electrophysiology examination without facial paralysis
5. patients with preoperative electrical testing without hearing impairment

Exclusion Criteria:

1. patients with poor compliance;
2. major surgical complications and interruption of treatment;
3. brain magnetic resonance examination or blood test results abnormal and clinical significance;
4. clinical trials of other drugs within 30 days;
5. the unintended side effects;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
House-Brackmann facial nerve grading scale | up to 3 months

IPD SHARING:
Plan to Share IPD: Yes